CLINICAL TRIAL: NCT06645626
Title: Utilisation of Health Services and Quality of Life in Patients With Atypical Parkinsonian Syndromes
Acronym: UHSQOLAPS
Status: Recruiting | Type: Observational
Sponsor: University Hospital Southampton NHS Foundation Trust (Other)
Responsible Party: Sponsor
Other Study IDs: NEU0416
Record Dates: First submitted 2022-09-30; First posted 2024-10-17 (Actual); Last update posted 2024-10-17 (Actual); Status verified 2024-10

CONDITIONS: Progressive Supranuclear Palsy; Cortico Basal Degeneration; Multiple System Atrophy
Keywords: quality of life; health economics
MeSH Terms: conditions — Supranuclear Palsy, Progressive; Corticobasal Degeneration; Multiple System Atrophy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- UHS Specialist Clinic population: All patients seen in regional clinic with this diagnosis
- Interested patients from non-specialty clinics around the country.: Interested patients who meet the inclusion criteria and are from any region in the country with no movement disorder specialist clinic.

SUMMARY:
The study will compare health care utilisation and quality of life for patients with progressive supranuclear palsy, corticobasal syndrome and multiple system atrophy in different parts of the region that our specialist clinic operates in with different services as well as in other regions with no specialist clinics. This study aims to investigate which aspects of the service are most beneficial for the patients and to determine the influence of support services and specialty clinics on patients and their carers.

DETAILED DESCRIPTION:
Progressive supranuclear palsy (PSP), Multiple system atrophy (MSA) and corticobasal syndrome (CBS) are rare neurological diseases which rapidly get worse. They cause problems with movement, vision, thinking, swallowing and speech and currently have no treatment to cure the disease or to treat many of the symptoms. They look superficially like Parkinson's disease and so are called collectively atypical Parkinsonian syndromes (APS). Quality of life for patients and their family is very poor; worse than motor neuron disease for example. Due to all the problems related to their illness patients often have to be admitted as an emergency and need a lot of care. Currently there is little research on how patients should be cared for by the NHS. While there are many variations in types of clinics, two different models for NHS clinics are 1) a Neurology Consultant seeing them in clinic alone or 2) a Neurologist seeing them in a specialist multidisciplinary (MDT) clinic with a clinic coordinator in close cooperation with community teams consisting of speech and language therapists, physiotherapists, occupational therapists, palliative care and a Neurology nurse. The second type of clinic would be more expensive but may provide the patient and their family with more information about the disease and support. This could improve the patient and carer's ability to manage the disease, the patient and carer's quality of life and experience of care, and may reduce emergency admissions to hospital. The clinic the investigators run in Wessex covers three counties with a wide variation in services on offer. In some of the patch community services are scarce and patients find it very difficult to come into the central clinic where the coordinator is based. In other parts there is a very comprehensive service with coordinators and multiple health professionals organised into a responsive and dedicated community MDT. The variation of MDT involvement in our clinic's catchment area enables us to study the influence of different levels of support on our patients.

Our study includes two stages: In the first stage, we will investigate the impact of different availability of services within our specialist clinic catchment area to determine the relative impact of support services on patients and their carers. The second stage will compare patients from our specialist clinic to patients seen elsewhere in the country in a non specialist setting. This will provide a much starker contrast of differences in care and outcomes.

Patient recruitment would be from our clinic list; however for patients who do not attend a specialist centre from different regions of the country we will be collaborating with the PSP Association (PSPA) to help us identify interested patients.

Informed consent is an absolute pre-requisite for participation in this study. Explicit consent will be obtained at the start of the study with regards ongoing involvement in the study in the event of loss of capacity. This research will assess patients using quantitative methods. Using questionnaires, patients and their carers (i.e. family members or friends who provide unpaid support) will be asked about their quality of life and how much the patients use health services at the beginning of the research and every 6 months to see if there is a difference between the types of care.

Quality of life data will be collected using a commonly used (EQ-5D-5L) or disease specific (PQOL, PSPQOL, MSAQOL) QOL measures. Additional information will be collected from patients including age, disease duration, medication, impulsivity & apathy (collected using the Cambridge Behavioural inventory revised [CBI-r] and the Cambridge Questionnaire for Apathy and Impulsivity Traits [CAMQUAIT - A Cambridge questionnaire).

Disease severity and cognition will be assessed using Montreal Cognitive Assessment [MOCA] for cognition and PSP rating scale [PSPRS], PSP Clinical Deficits scale[PSPCDS] or unified MSA rating scale [UMSARS] for disease severity to ensure that recruited patients are as similar as possible with regard to disease type, stage and disability. The researcher will also access clinical data to provide contextual information regarding the patient and their disease as outlined above. This will predominantly be at UHS for QOLAPS1 patients but may also be requested from other hospitals in the region and the GP. For QOLAPS2 patients we will request information from any NHS hospital in the region and their GP. We will also request data from NHS digital and other UK NHS databases - in particular the Office of National Statistics (ONS). This will predominantly be for mortality data which will enable us to look at outcomes including duration of disease, cause and place of death and we will look to relate that to the clinical care patients received.

A few of the assessments require an in-person assessment such as the MOCA and the PSPRS, PSPCDS or UMSARS. These measures are often a normal part of our clinical care and will be done at the patient's clinic visit. For the group of patients who are not attending our clinics, we would arrange a home visit and carry out the assessments at the patient's home.

ELIGIBILITY:
Inclusion Criteria:

Patients and their carers must:

* Be aged 18 or over
* Have capacity to consent at the beginning of their involvement
* Have a diagnosis of a neurodegenerative disease which includes progressive supranuclear palsy, corticobasal syndrome and multiple system atrophy but may include other closely related diseases where the presentation is similar, such as Alzheimer's disease where they present with a corticobasal syndrome

Exclusion Criteria:

* Patients or carers not meeting the inclusion criteria
* Patients with static deficits only who do not have a neurodegenerative syndrome.
* Patients who the principal investigator feels are not suitable to take part due to co-morbidities or participation in other trials.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients attending the Wessex Atypical Parkinsonian syndrome clinic. Patients not attending the Wessex Atypical Parkinsonian syndrome clinic or any movement disorder specialist clinic in the UK.
Sampling Method: Non-Probability Sample
Enrollment: 198 (Estimated)
Dates: Start 2022-10-10 (Actual); Primary Completion 2026-08-31 (Estimated); Study Completion 2027-07-15 (Estimated)

PRIMARY OUTCOMES:
Change in Quality of life score | Change in quality of life score from enrolment to 12 months of participation
  Quality of life assessments using disease specific measures: the progressive supranuclear syndrome quality of life scale (Minimum score 0 and Max (worst) score is 180), Multiple system atrophy quality of life scale (minimum (best) score 0 and maximum score (worst) 160) and generic scales: the EQ5D5L (minimum (best) 0 and maximum (worst) 20) for patients and carers.
Change in health utilisation cost | Change in health utilisation cost from enrolment to 12 months of participation
  Cost to the health service using the Resource utilisation in Dementia scale.

SECONDARY OUTCOMES:
Time to disease milestones | Assessment of patients function from baseline at the time of enrolment to 12 months of participation
  Time between onset of symptoms to assistance with walking, use of wheelchair, urinary catheter, nursing home and death. Better outcomes would be delayed time to disease milestones.

CONTACTS AND LOCATIONS:
Overall Officials: Boyd CP Ghosh, MBBS, Principal Investigator — Wessex Neurological Centre
Locations (1):
- Wessex Neurological Centre, Southampton, Hampshire, United Kingdom

IPD SHARING:
Plan to Share IPD: No
No current plans